CLINICAL TRIAL: NCT06395584
Title: Analysis of the Central Pathways Responsible for Green Light Therapy-Induced Pain Relief in Osteoarthritis
Brief Title: Light Therapy and MRI Imaging for Knee Osteoarthritis Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63924
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups: one group will receive daily light therapy treatments and the second group will not.
Who Masked: Participant
Masking Description: Participants assigned to the light therapy treatment group will use two different colours of light (white and green). One colour is a treatment light and the other is a placebo. Participants will not be told which is the treatment colour and which is the placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light therapy group (Active Comparator): Participants will be asked to use two different colours of light for 1-2 hours/day in a dark room in their home for 20 weeks. They will first use a white light for 10 weeks, followed by a green light for 10 weeks. They will be asked to complete daily pain diaries and a series of 3 MRI brain scans.
  Interventions: Device: White Light LED; Device: Green Light LED
- No light therapy group (No Intervention): Participants will not receive light intervention but will be asked to complete daily pain diaries and a series of 3 MRI brain scans.

INTERVENTIONS:
Device: White Light LED — Participants will be exposed to white LED lights (4 lux) in a dark room for 1-2 hours per day for 10 weeks.
  Arms: Light therapy group
Device: Green Light LED — Participants will be exposed to green LED lights (4 lux) in a dark room for 1-2 hours per day for 10 weeks.
  Arms: Light therapy group

SUMMARY:
Managing joint pain is one of the main goals for treating osteoarthritis (OA) and other musculoskeletal disorders. Alleviating chronic pain pharmacologically has several potential drawbacks including diminishing efficacy, toxicity, adverse side-effects, and patient anxiety. Non-pharmacological approaches (eg. weight loss) have also been found to be effective at controlling joint pain and can provide supplementary benefits. The development of efficacious, alternative treatments for arthritis pain which provide analgesia without adverse side-effects would be advantageous.

Recently, preclinical and clinical studies have demonstrated that green ambient light using light-emitting diodes (LEDs) produced profound analgesia in animal models and chronic pain patients. Both migraineurs and fibromyalgia patients have both reported significant reductions in pain following 10 weeks of green LED exposure.

It is unknown how green light reduces pain, but it is believed to be in the connections between the visual and pain control centres in the brain. Investigators will examine whether green light reduces OA knee pain by altering pain processes in the brain. To assess this, we will recruit 44 participants and randomly assign them to one of two groups: one group will receive light treatments every day for 20 weeks and the other group will not. We will ask both groups to report pain in daily pain diaries and ask both groups to have a series of 3 MRI brain scans to determine if light exposure changes how the brain processes pain.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis, yet treatment options are limited to pain management. Non-steroidal anti-inflammatory drugs (NSAIDs) and corticosteroids are the pharmacological foundation of OA pain control; however, prolonged use can come with considerable potential side effects that compromise (among others) heart, liver, and bone health. Thus, alternative non-pharmacological treatments may prove beneficial for a safe and more desirable alleviation of arthritis pain.

Recent preclinical and clinical studies discovered that viewing dim green ambient light for 1-2 hours per day for 10 weeks dramatically reduced pain levels. Using light-emitting diodes, migraineurs exposed to this green light therapy (GLT) reported a significant reduction in both headache days as well as headache intensity. Treating the same study participants with white light as a control had no effect on reported pain levels indicating that light specifically in the green range was necessary for analgesia. Critically, exposure to these low intensity light-emitting diodes produced no adverse side-effects and was easily tolerated by patients.

A pre-clinical study of rodents revealed that exposure to green light reduced joint pain in a rat model of OA and this effect was mediated in part by the endocannabinoid system. The mechanism by which green light produces analgesia is unknown, but there is believed to be neural connections between the visual system and pain control centres in the brain. Endogenous opioid release and descending inhibitory pathways are also believed to be involved in GLT responses. Whether green light alleviates OA pain by altering pain processes in the central nervous system has not been investigated. Therefore, the hypothesis to be tested in this project is: The analgesic effect of green light therapy in OA is mediated by central inhibitory pain circuits.

The primary specific aim of this project is to examine changes in brain circuitry in patients with OA following green light therapy. We will achieve this by recruiting 44 participants with knee OA and randomly assigning them to an active group or a control group. The active group will first receive a daily placebo (white) light intervention for 10 weeks, followed by a daily treatment (green) light intervention for 10 weeks. Participants will be asked to participate in brain imaging scans at baseline and then following white light intervention and green light interventions. The control group will receive no light intervention but will be asked to participate in time-matched fMRI scans. fMRI data will be compared between the active and control groups. We will also ask participants in both groups to self-report measures of knee pain and functioning throughout the study using various questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee
* 18 years of age or older
* Right-handedness
* Stable pain medication use during the previous 14 days
* At least 4/10 knee pain, on average during the previous 14 days
* Able to get onto an MRI table with minimal support
* Comfortable completing questionnaires and study tasks with English language instructions

Exclusion Criteria:

* Visual impairments that cannot be corrected using prescription glasses or contact lenses
* Currently enrolled in other clinical trial involving a pharmaceutical treatment
* Knee surgery scheduled within 8 months of study initiation
* History of cardiac, respiratory, or nervous system disease that may interfere with participation in the study or cause heightened potential for adverse outcome. For example: asthma or claustrophobia
* Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score Diary | 24 weeks
  Change in mean daily pain diary score from baseline (average pain score over 7 days pre-treatment) to post treatment

SECONDARY OUTCOMES:
The Western Ontario and McMaster University Arthritis Index | 24 weeks
  Change in WOMAC score from baseline to post treatments
The Brief Pain Inventory Short Form | 24 weeks
  Change in BPI score from baseline to post treatments
The Global Impression of Change and Satisfaction | 24 weeks
  Change to quality of life will be assessed post treatments
The Pain Catastrophizing Scale | 24 weeks
  Change in PCS score from baseline to post treatments
Five Facet Mindfulness Questionnaire | 24 weeks
  Change in FFMQ score from baseline to post treatments
The Spielberger Trait Anxiety Inventory | 24 weeks
  Change in STAI score from baseline to post treatments
Pain vigilance questionnaire | 24 weeks
  Change in PVAQ score from baseline to post treatments
Medication Quantification Scale | 24 weeks
  Change in MQS score from baseline to post treatments

OTHER OUTCOMES:
fMRI brain scans | 24 weeks
  Examination of brain scans taken at baseline and (2) post treatments

CONTACTS AND LOCATIONS:
Overall Officials: Karim Mukhida, MD, PhD, Principal Investigator — NS Health
Locations (1):
- NS Health, Halifax, Nova Scotia, Canada